CLINICAL TRIAL: NCT04288856
Title: An Extension Study to Assess the Long-Term Safety, Tolerability, Pharmacokinetics, and Effect on Disease Progression of BIIB078 Administered to Previously Treated Adults With C9ORF72-Associated Amyotrophic Lateral Sclerosis
Brief Title: Study to Assess the Safety, Tolerability, Pharmacokinetics, and Effect on Disease Progression of BIIB078 Administered to Previously Treated Adults C9ORF72-Associated Amyotrophic Lateral Sclerosis (ALS)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: There was no evidence of benefit across efficacy endpoints in the randomized trial, 245AS101. Accordingly, Biogen has made the difficult decision to discontinue the BIIB078 program including this open label extension trial, 245AS102.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 245AS102; 2019-004798-14 (EudraCT Number)
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Masking Description: During the blinded loading period, the following individuals will be masked:
  * Investigator
  * Study staff
  * Participants
  After the loading period has been completed, subsequent doses will be open-label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A: BIIB078 First Dosage (Experimental): BIIB078 will be administered as 3 doses during the loading period, approximately 2 weeks apart, and maintenance doses, approximately 4 weeks apart, via IT infusion.
  Interventions: Drug: BIIB078
- Cohort B: BIIB078 Second Dosage (Experimental): BIIB078 will be administered as 3 doses during the loading period, approximately 2 weeks apart, and maintenance doses, approximately 4 weeks apart, via IT infusion.
  Interventions: Drug: BIIB078
- Cohort C: BIIB078 Third Dosage (Experimental): BIIB078 will be administered as 3 doses during the loading period, approximately 2 weeks apart, and maintenance doses, approximately 4 weeks apart, via IT infusion.
  Interventions: Drug: BIIB078
- Possible Cohort D: BIIB078 Fourth Dosage (Experimental): BIIB078 will be administered as 3 doses during the loading period, approximately 2 weeks apart, and maintenance doses, approximately 4 weeks apart, via IT infusion.
  Interventions: Drug: BIIB078

INTERVENTIONS:
Drug: BIIB078 — Administered as specified in the treatment arm.

SUMMARY:
The primary objective is to evaluate the long-term safety and tolerability of BIIB078 in participants with chromosome 9 open reading frame 72-amyotrophic lateral sclerosis (C9ORF72-ALS).

The secondary objective is to evaluate the pharmacokinectic (PK) of BIIB078 in participants with C9ORF72-ALS.

DETAILED DESCRIPTION:
This study is an extension study of NCT03626012.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must have completed study NCT03626012 through the first follow-up clinic visit that follows the final dosing visit without missing more than 1 dose of study treatment.
* Participants taking concomitant riluzole at study entry must be on a stable dose for ≥30 days prior to the first dose of study treatment (Day 1). Participants taking concomitant riluzole must be willing to continue with the same dose regimen throughout the study, unless the Investigator determines that riluzole should be discontinued for medical reasons, in which case it may not be restarted during the study.
* Participants taking concomitant edaravone at study entry must be on a stable dose for ≥60 days prior to the first dose of study treatment (Day 1). Participants taking concomitant edaravone must be willing to continue with the same dose regimen throughout the study, unless the Investigator determines that edaravone should be discontinued for medical reasons, in which case it may not be restarted during the study. Edaravone may not be administered on dosing days of this study.

Key Exclusion Criteria:

* History of drug abuse or alcoholism ≤6 months before study enrollment that would limit participation in the study, as determined by the Investigator.
* Presence of an implanted shunt for the drainage of CSF or an implanted central nervous system (CNS) catheter.
* History of or positive test result at Screening for human immunodeficiency virus. The requirement for testing at Screening may be omitted if it is not permitted by local regulations.
* Treatment with another investigational drug (including investigational drugs for ALS through compassionate use programs) or biological agent within 1 month of Screening or 5 half-lives of study agent, whichever is longer.

Note: Other protocol-specific inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Baseline up to Day 785
  AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Number of Participants with Serious Adverse Events (SAEs) | Screening up to Day 785
  An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment.

SECONDARY OUTCOMES:
Serum concentration of BIIB078 | Baseline and at multiple time points up to Day 729
Cerebrospinal Fluid (CSF) concentration of BIIB078 | Baseline and at multiple time points up to Day 729

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (20):
- United States (12):
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, Palo Alto, California
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, New York, New York
  - Research Site, Knoxville, Tennessee
- Canada (4):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Research Site, Utrecht, Netherlands
- Research Site, Sankt Gallen, Switzerland
- United Kingdom (2):
  - Research Site, London, Greater London
  - Research Site, Sheffield, South Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/